CLINICAL TRIAL: NCT01074385
Title: Use of Dignity Therapy in Stage IV Colorectal Cancer Patients Receiving Chemotherapy to Increase Peaceful Awareness and Impact Goals of Care Decision-Making
Brief Title: Dignity Therapy in mCRC to Increase Peaceful Awareness & Impact Goals of Care Decision-Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NU 09CC3; STU00022908 (Other: Northwestern University IRB); NCI-2010-01851 (Other: NCI CTRP#)
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Stage IV Colorectal Cancer
Keywords: Stage IV Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Dignity Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Dignity Therapy (Other): At registration, subjects will be mailed a questionnaire. The subject will then receive two separate dignity therapy sessions, about a week apart. Subjects will then be asked to complete a questionnaire 1-2 weeks after completing therapy sessions and one month after completing therapy sessions.
  Interventions: Behavioral: Dignity Therapy
- Wait List Dignity Therapy (Other): At registration, subjects will be mailed a questionnaire. The subject will then receive two separate dignity therapy sessions; the first session will take place about 6 weeks after registration, with the second session occurring 1-3 weeks after the first. Subjects will then be asked to complete a questionnaire about one month after completing therapy sessions.
  Interventions: Behavioral: Dignity Therapy

INTERVENTIONS:
Behavioral: Dignity Therapy — Dignity therapy is a psychotherapeutic intervention developed to address psychosocial and existential distress among terminally ill patients. Basically, it invites patients to discuss topics that matter most or how they want to be remembered. This interview is recorded and then edited and returned to the patient to be used for further reflection or for sharing with loved ones.

SUMMARY:
The purpose of this study is to try and improve the way that patients with colon cancer understand and cope with their illness and give them tools for talking with their loved ones and family about their illness.

DETAILED DESCRIPTION:
Dignity Therapy is a well tolerated structured interview that helps patients reflect on who they are, what is most important to them and what lessons they have learned through life. For patients not receiving chemotherapy, Dignity Therapy gave patients more hope, more meaning in their life, and helped their families. Researchers at Northwestern University would like to see if it has the same effect in patients getting chemotherapy. We will also see if the Dignity Therapy changes patient's understanding of their disease and their medical preferences.

All study procedures will take place when participants come for a scheduled doctor's visit or to receive chemotherapy. At the first visit participants will answer a questionnaire taking approximately 15-30 minutes. Participants will then have a Dignity Therapy Session approximately 1-2 weeks later. A second Dignity Therapy Session will be scheduled again in another 1-2 weeks. Each study Dignity Therapy Session will take approximately an hour. One to two weeks later a repeat questionnaire will be filled out. Finally, a third and final questionnaire will be complete 4 weeks later.

ELIGIBILITY:
* Participants must be currently receiving treatment for stage IV colorectal cancer.
* Participants must have experience disease progression after their first course of treatment and are being considered for second course of treatment or have already started their second course of treatment.
* Participants must be 18 years old or older.
* All participants must have given signed, informed consent prior to registration on study.
* Participants must speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Impact of Dignity Therapy | at baseline, 1-2 weeks after completion of dignity therapy sessions, 1 month after completion of sessions
  Measure the impact of dignity therapy on terminal illness acknowledgment and presence of peaceful awareness. Subjects will complete self-evaluation questionnaires at the point of registration and upon completing dignity therapy sessions. The impact will be determined by changes in the patient's baseline self-reported parameters.

SECONDARY OUTCOMES:
Measure the impact of dignity therapy on life sustaining therapy and end-of-life goals of care. | at baseline, 1-2 weeks after completion of dignity therapy sessions, 1 month after completion of dignity therapy sessions
  Subjects will complete self-evaluation questionnaires at the point of registration and upon completing dignity therapy sessions. The impact will be determined by changes in the patient's baseline self-reported parameters.
Establish a correlation between terminal illness acknowledgement and presence of peaceful awareness with preferences for life sustaining therapy and end-of-life goals of care. | At Study Completion
  Establish a correlation between terminal illness acknowledgement and presence of peaceful awareness with preferences for life sustaining therapy and end-of-life goals of care.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Emanuel, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Northwestern Memorial Faculty Foundation, Chicago, Illinois, United States